CLINICAL TRIAL: NCT06345469
Title: Cost Effectiveness Analysis of Transfusion Therapy and Patient Blood Management in Patients With Severe Anemia
Brief Title: Cost Analysis of Therapies for Severe Anemia
Status: Not yet recruiting | Type: Observational
Sponsor: Helios Klinik Gotha/Ohrdruf (Other)
Collaborators: Marisa Eichner (Unknown)
Responsible Party: Principal Investigator, Petra Seeber, Principal Investigator, Helios Klinik Gotha/Ohrdruf
Other Study IDs: O-PBM2
Record Dates: First submitted 2024-03-25; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Severe Anemia
Keywords: anemia; costs; transfusion; patient blood management
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PBM only: The Study group received comprehensive Patient Blood Management without allogeneic transfusions to treat their severe anemia.
  Interventions: Other: Patient blood management (PBM)
- PBM with transfusion: The Control group opted to be treated with allogeneic transfusions together with convenience measures of PBM.
  Interventions: Other: Patient blood management (PBM); Biological: Allogeneic transfusion

INTERVENTIONS:
Other: Patient blood management (PBM) — PBM means the medical enhancement of the participants own hematopoietic reserve to treat anemia and to reduce the ill effects of disease and bleeding on hematopoiesis and homeostasis.
Biological: Allogeneic transfusion — transfusion of donor red cells
  Groups: PBM with transfusion

SUMMARY:
The goal of this observational study is to learn about the costs that occur when participants with severe anemia are treated with blood transfusions or with patient blood management (PBM). PBM means that the body of the participant is stimulated to produce new blood by itself rather than receiving it from a blood donor, and to reduce blood losses.

The main question the study aims to answer is: Do participants treated with transfusions incur the same treatment costs than participants treated with PBM? And how much costs are this in relation to the lives saved by the therapy of severe anemia?

DETAILED DESCRIPTION:
Background:

Severe anemia is a condition that is associated with increased morbidity and mortality in hospitalized patients. In an effort to treat severe anemia, transfusions and/or Patient Blood Management are provided with the goal to reduce morbidity and mortality. This treatment naturally incurs costs. Several studies already tried to evaluate the costs of transfusions and PBM and to compare them. However, a comparison of the therapy costs of severe anemia and their cost effectiveness is not available.

Objective: It is the objective of this study to assess therapeutic costs of severe anemia and to compare the cost effectiveness of transfusion therapy and PBM in relation to their effect on inhospital mortality.

Hypothesis: It is hypothesized that the therapy of severely anemic participants who received PBM and who receive transfusions is equally cost effective as regards its ability to reduce in-hospital mortality.

Setting: The study will be performed at HELIOS Klinikum Gotha, a hospital with general, advanced and specialized care which offers not only transfusions but also PBM.

Data sources: Data will be sourced from the hospital information system as well as from chart review.

Participants: All adult patients treated between 2008 and 2020 in Helios Klinikum Gotha who had a nadir hemoglobin of less than 8 g/dL and who opted to be treated with PBM, but not with allogeneic transfusions. A control group will be matched from all other severely anemic patients treated in the same time period but who opted to receive transfusions.

Interventions: allogeneic transfusion therapy with red blood cells according to the standards of the Federal Chamber of Physicians in Germany or Patient Blood Management only without transfusion of allogeneic red cells.

Outcome:

The primary outcome is the cost-effectiveness of transfusion therapy and PBM to reduce in-hospital mortality.

Costs will be calculated by the top-down and the bottom-up method and the Incremental Cost Effectiveness Ratio (ICER) will be calculated in relation to mortality reduction.

Study design:

This is a retrospective observational cohort study. Reporting of the results will be performed in line with the CHEERS (Consolidated Health Economic Evaluation Reporting Standards 2022) statement.

The study will be guided by a study protocol with an attached statistical analysis plan.

ELIGIBILITY:
Inclusion Criteria:

* adult (> 18 years at admission)
* hemoglobin nadir of < 8 g/dL

Exclusion Criteria:

* participants treated by physicians not related to Helios Klinikum Gotha

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants admitted to Helios Klinikum Gotha, Germany, between 2008 and 2020
Sampling Method: Probability Sample
Enrollment: 640 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
cost-effectiveness | From date of admission to hospital until the date of discharge or date of death from any cause, whichever came first, assessed for the whole hospitalization period, assessed up to 100 months
  The study evaluates costs incurred to treat severe anemia and how these relates to its effect on reduction of inhospital mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Petra Seeber, MD, Principal Investigator — HELIOS Klinikum Gotha

IPD SHARING:
Plan to Share IPD: No